CLINICAL TRIAL: NCT05045508
Title: A Randomized, Controlled, Double-Masked, Two-Arm Investigator-Initiated Study to Assess the Efficacy of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease Following Photorefractive Keratectomy (PRK)
Brief Title: Investigator Initiated Study to Assess the Efficacy of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease Following Photorefractive Keratectomy (PRK)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brandon Baartman (Other)
Responsible Party: Sponsor-Investigator, Brandon Baartman, Brandon Baartman, Principal Investigator, Vance Thompson Vision NE
Organization: Vance Thompson Vision NE (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: The MyOpe Study
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC-01 (varenicline 0.6mg/ml) nasal spray (Experimental)
  Interventions: Drug: OC-01 (varenicline 0.6mg/ml) nasal spray
- Placebo (vehicle) nasal spray (Placebo Comparator)
  Interventions: Drug: Placebo (vehicle) Nasal Spray

INTERVENTIONS:
Drug: OC-01 (varenicline 0.6mg/ml) nasal spray — OC-01 nasal spray which contains varenicline is being developed by Oyster Point Pharma for the treatment of signs and symptoms of DED. OC-01 (varenicline) nasal spray activates the trigeminal parasympathetic pathway and stimulates natural tear production and bathe the corneal nerve endings in a protective layer of tear film. In addition, OC-01 (varenicline) acts as a cholinergic agonist and may provide analgesia by activating the trigeminal parasympathetic pathway.
  Arms: OC-01 (varenicline 0.6mg/ml) nasal spray
Drug: Placebo (vehicle) Nasal Spray — Placebo (vehicle) nasal spray [control]
  Arms: Placebo (vehicle) nasal spray

SUMMARY:
Evaluate the safety and effectiveness of OC-01 (varenicline) nasal spray among subjects suffering from dry eye following photorefractive keratectomy (PRK)

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign the informed consent form (ICF)
* Be at least 18 years of age at the screening visit
* Be undergoing PRK treatment in one or both eyes
* Be myopic between -1.00D to 6.00D manifest refraction spherical equivalent (MRSE) in study eye (right eye) with ≤2D between eyes or subjects undergoing monovision treatment with study eye being the distance eye and meeting the MRSE requirement of myopia
* Be literate and able to complete questionnaires independently
* Be able and willing to use the study drug and participate in all study assessments and visits
* Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug
* Have provided written informed consent
* If a female is of childbearing potential, they must: use an acceptable means of birth control (acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives, mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom, IUD, or surgical sterilization of partner), and have a negative urine pregnancy test on baseline visit and form of birth control will be documented

Exclusion Criteria:

Have a break in the integrity of the corneal epithelium such as a persistent corneal epithelial defect or corneal ulcer.

* Have placement of temporary punctal plugs in the past 1 month or current presence of permanent punctal plugs at time of screening
* Presence of corneal pathology that may interfere with PRK outcomes Active infectious, ocular or systemic disease
* Patients with a history of ocular inflammation or macular edema
* Clinically significant active infectious keratitis in the past 3 months
* Have had prior refractive surgery
* Have chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to clinically significant risk of increased bleeding
* Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Have a vascularized polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal obstruction as confirmed by intranasal examination performed at Visit 1.
* Be currently treated with nasal continuous positive airway pressure
* Have had blepharoplasty in either eye
* Have had a corneal transplant in either eye
* Have a history of seizures or other factors that lower the subject's seizure threshold.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have current concomitant use of a nicotinic acetylcholine receptor agonist [Nicoderm®, Nicorette®, Nicotrol NS® (nicotine), Tabex®, Desmoxan® (cytisine), and Chantix® (varenicline)] within the previous 30 days of Visit 1 and during the treatment period.
* Have active or uncontrolled, severe at the discretion of the investigator:

  * Systemic allergy
  * Chronic seasonal allergies at risk of being active during the study treatment period
  * Rhinitis or sinusitis requiring treatment such as antihistamines, decongestants, oral or aerosol steroids at the Screening Visit or be expected to require treatment during the treatment period of the study
* Have untreated nasal infection at Visit 1
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1 and during the treatment period.
* Be a female who is pregnant, nursing, or planning a pregnancy at Visit 1. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire) score | From baseline to day 84 (3 months)
  25 questions to determine overall score of dry eye disease symptoms completed by subject
Change in corneal epithelial healing | from 2 days (48hours) post op to 7 days (1 week) post op
  evaluated at the slit lamp by a masked physician

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Baartman, MD, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Omaha, Nebraska, United States